CLINICAL TRIAL: NCT05886036
Title: NORM: Nodular Lymphocyte-Predominant Hodgkin Lymphoma Patients Treated in a Randomized Phase 2 Trial With Either Rituximab or Mosunetuzumab
Brief Title: Comparing the Effectiveness of the Immunotherapy Agents Rituximab or Mosunetuzumab in Patients With Nodular Lymphocyte-Predominant Hodgkin Lymphoma, NORM Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-04108; NCI-2023-04108 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10590 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10590 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2023-06-01; First posted 2023-06-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Nodular Lymphocyte Predominant B-Cell Lymphoma; Recurrent Nodular Lymphocyte Predominant B-Cell Lymphoma; Refractory Nodular Lymphocyte Predominant B-Cell Lymphoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Rituximab; CT-P10; Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Mosunetuzumab) (Experimental): Patients receive mosunetuzumab SC on days 1, 8, and 15 of cycle 1 and day 1 of subsequent cycles. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients who experience PD will be permitted to crossover to arm II at week 12. Patients also receive FDG and undergo PET/CT at baseline and end of treatment. Patients who are positive at pre-treatment bone marrow biopsy also receive FDG and undergo PET/CT on study. Patients also undergo bone marrow biopsy and tissue biopsy at baseline, and blood sample collection throughout the trial. Patients may also undergo bone marrow biopsy and tissue biopsy at end of treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Biological: Mosunetuzumab; Procedure: Positron Emission Tomography
- Arm II (Rituximab, Rituximab and hyaluronidase human) (Active Comparator): Patients receive rituximab IV on day 1 and rituximab and hyaluronidase human SC on days 8, 15, and 22 of each cycle. Cycles repeat every 28 days for up to 2 cycles 8 weeks apart in the absence of disease progression or unacceptable toxicity. Patients may receive rituximab IV on days 8, 15, and 22 of each cycle if rituximab and hyaluronidase human is not available. Patients who experience PD will be permitted to crossover to arm I at week 12. Patients also receive FDG and undergo PET/CT at baseline and end of treatment. Patients who are positive at pre-treatment bone marrow biopsy also receive FDG and undergo PET/CT on study. Patients also undergo bone marrow biopsy and tissue biopsy at baseline, and blood sample collection throughout the trial. Patients may also undergo bone marrow biopsy and tissue biopsy at end of treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Fludeoxyglucose F-18 — Receive FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Biological: Mosunetuzumab — Given SC
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody BTCT4465A; BTCT 4465A; BTCT-4465A; BTCT4465A; CD20/CD3 BiMAb BTCT4465A; Lunsumio; Mosunetuzumab-axgb; RG 7828; RG-7828; RG7828; RO7030816
  Arms: Arm I (Mosunetuzumab)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
  Arms: Arm II (Rituximab, Rituximab and hyaluronidase human)
Biological: Rituximab and Hyaluronidase Human — Given SC
  Other Names: Rituxan Hycela; Rituximab Plus Hyaluronidase; Rituximab/Hyaluronidase; Rituximab/Hyaluronidase Human
  Arms: Arm II (Rituximab, Rituximab and hyaluronidase human)

SUMMARY:
This phase II trial compares mosunetuzumab to the usual treatment (rituximab) for improving survival in patients with nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL). Rituximab and mosunetuzumab are monoclonal antibodies. They bind to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Mosunetuzumab may be more effective at extending survival in patients with NLPHL than the usual approach with rituximab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the progression-free survival (PFS) of mosunetuzumab versus rituximab in NLPHL patients.

SECONDARY OBJECTIVES:

I. To compare the safety and antitumor activity of NLPHL patients treated with mosunetuzumab versus rituximab.

II. To evaluate the molecular effects of mosunetuzumab and rituximab on tumor cells and the immune response and identify biomarkers of response or resistance with ribonucleic acid sequencing (RNAseq), whole exome sequencing (WES), immunohistochemistry (IHC) CD20, PD-1, PD-L1, PD-L2.

III. To evaluate tumor microenvironment and peripheral immune status with single-cell ribonucleic acid sequencing (scRNA-seq).

EXPLORATORY OBJECTIVES:

I. To evaluate CD20 expression and correlate with response. II. To evaluate the dynamic molecular response of NLPHL patients treated with rituximab or mosunetuzumab with circulating tumor deoxyribonucleic acid (ctDNA).

III. To evaluate the safety and efficacy (including tumor response, immune response, and overall survival) of the crossover patients.

IV. To assess the association of baseline fludeoxyglucose F-18 (FDG)-positron emission tomography/computed tomography (PET/CT) measurements including metabolic tumor volume (MTV) and maximum standardized uptake value (SUVmax), in combination with other risk factors, with PFS and overall survival (OS) in patients with lymphocyte-predominant Hodgkin lymphoma treated with mosunetuzumab or rituximab.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive mosunetuzumab subcutaneously (SC) on days 1, 8, and 15 of cycle 1 and day 1 of subsequent cycles. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients who experience progressive disease (PD) will be permitted to crossover to arm II at week 12. Patients also receive FDG and undergo PET/CT at baseline and end of treatment. Patients who are positive at pre-treatment bone marrow biopsy also receive FDG and undergo PET/CT on study. Patients also undergo bone marrow biopsy and tissue biopsy at baseline, and blood sample collection throughout the trial. Patients may also undergo bone marrow biopsy and tissue biopsy at end of treatment.

ARM II: Patients receive rituximab intravenously (IV) on day 1 and rituximab and hyaluronidase human SC on days 8, 15, and 22 of each cycle. Cycles repeat every 28 days for up to 2 cycles 8 weeks apart in the absence of disease progression or unacceptable toxicity. Patients may receive rituximab IV on days 8, 15, and 22 of each cycle if rituximab and hyaluronidase human is not available. Patients who experience PD will be permitted to crossover to arm I at week 12. Patients also receive FDG and undergo PET/CT at baseline and end of treatment. Patients who are positive at pre-treatment bone marrow biopsy also receive FDG and undergo PET/CT on study. Patients also undergo bone marrow biopsy and tissue biopsy at baseline, and blood sample collection throughout the trial. Patients may also undergo bone marrow biopsy and tissue biopsy at end of treatment.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of NLPHL as confirmed by local pathologist's expert review.

  * Untreated NLPHL: stage IB to IV according to Cotswolds. The proportion of patients with stages I or II treated with consolidative radiotherapy will be capped at 40%.
  * Previously treated NLPHL, any stage.
  * According to the treating physician, the patient should not be observed and needs therapy, notably because of B-symptoms (unexplained fever [temperature > 38 degrees Celsius (> 100.4 degrees Fahrenheit)], weight loss [unexplained loss of > 10 percent of body weight over the past six months], or drenching night sweats), symptomatic nodal or extranodal disease, or patient preferences.
* Patients must have measurable disease according to the Lugano/Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) classification.
* Age >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of mosunetuzumab in patients < 18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group performance status =< 2 (Karnofsky >= 60%).
* Absolute neutrophil count >= 1,000/mcL.
* Platelets >= 100,000/mcL.
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN), except in patients with Gilbert's syndrome as defined by > 80% unconjugated bilirubin.
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine transaminase (ALT)(serum glutamic-pyruvic transaminase [SGPT]) =< 3 x institutional ULN.
* Glomerular filtration rate (GFR) >= 40mL /min= GFR (mL/Min/1.73 m^2) * body surface area (BSA)/1.73.
* Human immunodeficiency virus-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* The effects of mosunetuzumab on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal and/or barrier method of birth control; abstinence) (both hormonal and barrier method of birth control are required for participants in Canada) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of mosunetuzumab administration and 12 months after completion of rituximab administration.
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Classical Hodgkin lymphoma (cHL) or composite lymphoma.
* Transformed NLPHL, concerns of the treating physician of an occult transformation or concerns of the treating physician that the patient needs cytotoxic therapy.
* NLPHL relapse less than 6 months after rituximab or rituximab-containing therapy.
* Patients who have not recovered from AEs due to prior anticancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* Patients with central nervous system (CNS) involvement as a result of lymphoma.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to mosunetuzumab or rituximab.
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous.
* Pregnant women are excluded from this study because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with mosunetuzumab; breastfeeding should be discontinued if the mother is treated with mosunetuzumab or rituximab. These potential risks may also apply to other agents used in this study.
* Prior allogeneic stem cell or solid organ transplantation.
* Participants who have received a live, attenuated vaccine within 4 weeks before first dose of study treatment or anticipation that such a live, attenuated vaccine will be required during the study. Participants must not receive live, attenuated vaccines (e.g., FluMist [registered trademark]) while receiving study treatment and after the last dose until B-cell recovery to the normal ranges. Killed vaccines or toxoids should be given at least 4 weeks prior to the first dose of study treatment to allow development of sufficient immunity.
* Any other anti-cancer therapy, whether investigational or approved, including but not limited to chemotherapy, within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to initiation of study treatment.
* Evidence of any significant, concomitant disease that could affect compliance with the protocol or interpretation of results as judged by the investigator, including, but not limited to:

  * Significant cardiovascular disease (e.g., New York Heart Association class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina).
  * Significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm).
  * Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease.
  * Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 1 year and have no residual neurologic deficits as judged by the investigator are allowed.
  * Participants with a history of epilepsy who have had no seizures in the past 2 years with or without anti-epileptic medications can be eligible only for the expansion cohort.
  * History of confirmed progressive multifocal leukoencephalopathy (PML).
* Participants with infections requiring IV treatment with antibiotics or hospitalization (grade 3 or 4) within the last 4 weeks prior to enrollment or known active bacterial, viral (including SARS-CoV-2), fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment.
* Systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to first dose of study treatment.
* Known or suspected chronic active Epstein-Barr virus (EBV) or cytomegalovirus (CMV) infection.
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) time | Time from the date of randomization to the first objective documentation of disease progression or death due to any cause, assessed up to 2 years
  Will be assessed according to the Lugano/Lymphoma Response to Immunomodulatory Therapy Criteria classification. The overall PFS curve will be displayed by treatment arm using the Kaplan-Meier (KM) method, and statistical comparisons will be performed by a log-rank test.

SECONDARY OUTCOMES:
Objective response | At week 12 and end of treatment
  The count and incidence rate of the response categories will be summarized for the overall population and by each treatment arm with a 95% exact confidence intervals. Comparison between treatment arms will be performed by a chi-squared test.
Duration of response | Time from the first date of partial or complete response until death or the assessment date of disease progression, assessed up to 2 years
  Will be displayed by treatment arm using the KM method, and statistical comparisons will be performed by a log-rank test.
Overall survival (OS) | Time from the date of randomization to death due to any cause, assessed up to 2 years
  Will be displayed by randomized treatment arm using the KM method, and statistical comparisons will be performed by a log-rank test.

OTHER OUTCOMES:
CD20 expression | Assessed up to 2 years
  CD20 expression will be evaluated and correlated with overall response rate, complete remission rate at end of treatment, and 2-year progression free survival.
Molecular effects of mosunetuzumab and rituximab on tumor cells and the immune response | Assessed up to 2 years
  Will assess the molecular effects of mosunetuzumab and rituximab on tumor cells and the immune response and identify biomarkers of response or resistance (objective response rate, complete remission rate at end of treatment, and 2-year PFS) with ribonucleic acid sequencing, whole exome sequencing, immunohistochemistry CD20, PD-1, PD-L1, and PD-L2.
Tumor microenvironment and peripheral immune status | Assessed up to 2 years
  Will be assessed by single-cell ribonucleic acid sequencing.
Dynamic molecular response of nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL) patients | During the first 7 weeks of treatment and at the end of treatment
  Will evaluate the dynamic molecular response of NLPHL patients treated with rituximab or mosunetuzumab with circulating tumor deoxyribonucleic acid.
Incidence of adverse events | Assessed up to 2 years
  Will be assessed by tumor response, immune response, and overall survival of the crossover patients.
Fludeoxyglucose F-18 positron emission tomography/computed tomography (FDG-PET/CT) measurements | At baseline
  Will assess the association of FDG-PET/CT measurements, including metabolic tumor volume and maximum standardized uptake value, in combination with other risk factors, with PFS and OS in patients with lymphocyte-predominant Hodgkin lymphoma treated with mosunetuzumab or rituximab.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael E Steiner, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (35):
- United States (34):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm